CLINICAL TRIAL: NCT04283318
Title: The Effects of Prolonged Fasting on Glucose Metabolism and Hormonal Regulation in Healthy, Obese and Subjects With Type 2 Diabetes
Brief Title: Prolonged Fasting on Glucose Metabolism and Hormonal Regulation in Healthy, Obese and Subjects With Type 2 Diabetes
Acronym: PROLOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HS-2018-01
Record Dates: First submitted 2019-02-18; First posted 2020-02-25 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Healthy; Obesity; Type 2 Diabetes Mellitus; Type 1 Diabetes
Keywords: starvation; healthy people; obese; Type 2 diabetes mellitus; glucose metabolism; Type 1 diabetes mellitus
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Starvation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy (Other): Age >18 years; BMI 20-27 kg/m2; Fasting plasma Glucose <110 mg/dL
  Interventions: Behavioral: 12h fasting; Behavioral: 36h fasting
- Obese people (Other): Age >18 years; BMI >30 kg/m2; Fasting Plasma Glucose <110 mg/dL
  Interventions: Behavioral: 12h fasting; Behavioral: 36h fasting
- Type 2 Diabetes (Other): Age >18 years; Diagnosed Type 2 Diabetes mellitus (diet or a monotherapy or combination of metformin, DPP-4-inhibitors or sulfonylurea)
  Interventions: Behavioral: 12h fasting; Behavioral: 36h fasting
- Type 1 Diabetes (Other): Age >18 years; Diagnosed Type 1 Diabetes mellitus >12 months; Treated with multiple daily Insulin injections (MDII) or continuous subcutaneous Insulin Infusion (CSII); Stable Insulin therapy as clinically assessed by the study physician C-Peptide negative defined as 0.3 nmol/L; No diabetic ketoacidosis within the last 12 months; No severe hypoglycaemia requiring external assistance within the last 12 months; Running on the FreeStyle Libre 1 (Abbott, USA) intermittently-viewed continuous Glucose Monitoring System (iCGM) as Standard of care for Glucose monitoring
  Interventions: Behavioral: 12h fasting; Behavioral: 36h fasting

INTERVENTIONS:
Behavioral: 12h fasting — 12h fasting (overnight)
Behavioral: 36h fasting — 36h fasting ( one day and two nights fasting)

SUMMARY:
In a previous study investigating the effects of intermittent fasting, our research group found evidence for higher glucose excursions and a reduced insulin response after a 36 hour fasting period as compared to an overnight fasting period in healthy subjects.

The aim of this research project is to investigate the effect of short and midterm fasting (12 hours versus 36 hours) on glucose metabolism, glucose regulatory hormones, insulin secretion and resting energy expenditure in healthy and obese people as well as in patients with type 2 diabetes.

DETAILED DESCRIPTION:
In this clinical study, we want to examine the effects of different fasting periods (12 hours versus 36 hours) on blood sugar levels and other metabolic parameters and hormones. For this the following investigations are carried out:

* Oral glucose tolerance test with detailed laboratory evaluation
* Bio-impedance measurement to determine body composition (muscle and fat mass)

The examinations are carried out on 4 different cohorts (normal healthy persons, obese patients, patients with type 2 diabetes and patients with type 1 diabetes).

ELIGIBILITY:
Gender: Both, male and female Minimum Age: 18 years

Inclusion Criteria Cohort I (Healthy, non-obese subjects) Age >18 years; body mass index in the range of 20.0-27.0 kg/m2; fasting plasma glucose <110mg/dL

Inclusion criteria cohort II (Obese subjects) Age >18 years; body mass index >30 kg/m2; fasting plasma glucose <110mg/dL

Inclusion Criteria Cohort III (Cohort with subjects with Type 2 Diabetes Mellitus) Age >18 years; established Diabetes mellitus type 2 on either diet or a monotherapy or combination of metformin, Dipeptidylpeptidase (DPP)-4-inhibitors or sulfonylurea

Inclusion Criteria Cohort IV (Cohort with subjects with Type 1 Diabetes Mellitus) Age >18 years; diagnosed with Type 1 Diabetes Mellitus >12 months; treated with multiple daily Insulin injectioins (MDII) or continuous subcutaneous Insulin Infusion (CSII); stable Insulin therapy as clinically assessed by the study physician; C-Peptide negative defined as 0.3 nmol/L; HbA1c <9.5%; no diabetic ketoacidosis within the last 12 months; no severe hypoglycaemia requiring external assistance within the last 12 months; running on the FreeStyle Libre 1 (Abbott, USA) intermittently-viewed continuous Glucose Monitoring System (iCGM) as Standard of care for Glucose monitoring

Exclusion Criteria (for all participants) History of cardiovascular disease; acute or chronic inflammatory disorder; heavy drinking (more than 15 drinks/week); dietary restrictions (e.g. vegetarianism and vegan); insulin Treatment (excluded subjects with Type 1 Diabetes Mellitus); corticosteroid therapy; known malignancy; women who are pregnant, breast-feeding or trying to become pregnant; history of any chronic disease process that could interfere with interpretation of study results; therapy with antidepressants within past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
change of 2h glucose levels | after 12 and 36 hours of fasting
  Difference in the change of 2h glucose levels in an oral glucose tolerance test

SECONDARY OUTCOMES:
changes in insulin sensitivity (QUICKI) | after 12 and 36 hours of fasting
  differences in QUICKI
changes in insulin sensitivity (Matsuda Index) | after 12 and 36 hours of fasting
  differences in Matsuda Index
changes in insulin sensitivity (ISI) | after 12 and 36 hours of fasting
  differences in ISI
changes in insulin sensitivity (HOMA-Index) | after 12 and 36 hours of fasting
  differences in HOMA-Index
Changes in glycaemic pattern | after 12 and 36 hours of fasting
  differences in area under the curve (AUC) of glycaemic pattern in Oral glucose tolerance test
Changes in body composition | after 12 and 36 hours of fasting
  differences in bioimpedance analysis

CONTACTS AND LOCATIONS:
Overall Officials: Harald Sourij, MD, Principal Investigator — Medical University of Graz, Auenbruggerplatz 15
Locations (1):
- Medical University of Graz, Graz, Austria